CLINICAL TRIAL: NCT04147741
Title: Effects of a Multi-Ingredient Pre-Workout on Performance, Perceptual Responses, Subjective Feelings of Energy and Muscular Contractile Properties, After a Resistance and Endurance Training Microcycle in Older Participants.
Brief Title: Effects of a Pre-Workout on Performance, Perceptual Responses, Energy Feelings and Muscular Properties, After a Training Microcycle in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Collaborators: Crown Sport Nutrition (Industry); Go Fit Spain (Unknown)
Responsible Party: Principal Investigator, Fernando Naclerio, Principal Lecturer, University of Greenwich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGreenwich
Record Dates: First submitted 2019-10-16; First posted 2019-11-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Protein Deficiency; Training Group, Sensitivity; Fatigue; Muscular Atrophy; Psychological
Keywords: Fatigue; Supplement; Pre-Workout; Muscle; Recovery; Training; Strength; Endurance; Perceptual Response
MeSH Terms: conditions — Protein Deficiency; Hypersensitivity; Fatigue; Muscular Atrophy | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Intervention Model Description: One week training (3 days Resistance Training and 2 Endurance Training in alternate days) with a Pre-Workout Supplement or Maltodextrin. 2 Weeks wash out period and then change supplement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Workout Supplement (Experimental): A 60 g dose of a commercially available pre-workout supplement providing 159 kcal including carbohydrates 15 g, essential amino acids 12 g, citrulline 3.5 g, Arginine, 3.5 g Taurine 1 g, L-Tyrosine 1 g, yerba mate 0.3 g and caffeine 0.4 g. With 250 ml of water.
  Interventions: Dietary Supplement: Pre-Workout Supplement; Other: Resistance Training; Other: Endurance Training
- Maltodextrin Supplement (Placebo Comparator): A isoenergetic Maltodextrin supplement will be administered as placebo. With 250 ml of water.
  Interventions: Dietary Supplement: Pre-Workout Supplement; Other: Resistance Training; Other: Endurance Training

INTERVENTIONS:
Dietary Supplement: Pre-Workout Supplement — One week familiarisation, one-week training, two weeks washout period and one-week training.
  15 Minutes before every training, the Pre-Workout Arm (PRE-W) will take a Supplement shake, consisting of some ingredients (Multi-Ingredient, explained before) and the Placebo Comparator Arm (CHO) will drink a Placebo shake, consisting of Maltodextrin.
  Other Names: Multi-Ingredient Supplement
Other: Resistance Training — -Resistance Training days (Monday-Wednesday-Friday): Before training starts, Tensiomyography and Energy Feeling will be assessed (Energy Level, Fatigue Level, Feeling of Alertness, and Feeling of Focus on the task). Immediately after finishing, Tensiomyography and Performance (Vertical Jump, Overhead Medicine Ball Throw, and Maximal Mid-Tigh Pull Isometric Strength) will be assessed. Training Protocol: 10 minutes of standardized warm-up, Strength Circuit training using free weights (Parallel Squat; Bench Press; Alternate Box Set-Ups; Shoulder Press; Alternate Lunges; Up-right Row; Hip-Thrust; Squat on Isoinertial Fly-Wheel or Drop Jump). The participants will have to perform 16 repetitions of each exercise, with 30 seconds rest and 3 minutes rest after every set. If they can complete 16 repetitions easily, 2,5 to 5 kg will be added for the next set. Also, whole-body Perceptual Response will be assessed using the 0-10 OMNI-RES Scale, after every set and 15 minutes after finishing.
  Other Names: Free Weights Training
Other: Endurance Training — - Endurance Training days (Tuesday-Thursday): Energy Feeling Questionnaire will be implemented before training. The training will consist of 30 minutes cycling at their Fatmax Intensity (~60% Vo2max) on a Cycloergometer (estimated during familiarisation week). Also, the Heart Rate will be recorded during the whole training. Besides, Perception of Effort will be assessed using the 6-20 version of the Borg Scale every 5 minutes during training and 15 minutes after it has been completed.
  Other Names: Cycloergometer Training

SUMMARY:
The investigation will be conducted as a double blinded, randomized, crossover within-participant comparison design with two 1-week intervention periods separated by 2-weeks for wash out, recovery, period.

DETAILED DESCRIPTION:
Following inclusion, familiarization and baseline assessments, the participants will be randomly allocated to receive either a multi-ingredient, pre-workout supplement (PREW) or maltodextrin (CHO). Thereafter, the participants will take a 5-day microcycle, involving three resistance training sessions (Monday, Wednesday and Friday) intercalated with two endurance training sessions (Tuesday and Thursday). After the first interventional microcycle, and the 2-week washout period, the participants will switch to the other nutritional condition for continuation with the second 5-day identical microcycle. Assessments of muscle contractile properties via Tensiomyography on Vastus Medialis, Biceps Femoris Long Head and Anterior Deltoids will be taken before and after each resistance training session. Measurements of strength (Isometric Mid Thigh Pull) upper and lower body muscular power (Medicine Ball Throw and Vertical Jump) will be performed immediately after each resistance training workout. The supplements will be ingested 15 min before each training session, just before completing an energy feeling questionnaire. In addition, the perceptual response to training will be assessed during and 20 min after the completion of all workouts. The contribution of carbohydrate and fat metabolism will be estimated using a gas analyzer via the calculation of respiratory exchange ratio the (RER) during each endurance training session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no current injuries).
* Between 45 and 70 years old.
* Active.

Exclusion Criteria:

* Injuries.
* Never trained before.
* Under 45 or over 70 years old.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Tensiomyography | Changes from 10 minutes Previous to post 1 hour after the completion of each workout session
  Fatigue and contractility assessment via Tensiomyography will be assessed in Biceps Femoris Long Head, Vastus Medialis, and Anterior Deltoid.
Vertical Jump | Changes from 10 minutes Previous to post 1 hour after the completion of each resistance training workout session
  Flight Time (measured in seconds).
Over Head Medicine Ball Throw | Changes from 10 minutes Previous to post 1 hour after the completion of each resistance training workout session
  Medicine Ball Throw (measured in meters and centimeters).
Maximal Mid-Thigh Pull Isometrical Strength | Changes from 10 minutes Previous to post 1 hour after the completion of each resistance training workout session
  Maximal Strength (measured in kilograms).
Self Perceived Energy Feeling | Before every Training Session and up to 1 week of training.
  All participants will fill a short questionnaire (from 1 to 5 points) about their perception of energy before every training.
  Energy Feeling will be assessed (Evergy level, Fatigue Level, Feeling of Alertness, and Feeling of Focus for the task, valued from 1 = low energy to 5 = high energy).

SECONDARY OUTCOMES:
Whole Body Perceptual Response during Resistance Training | Differences between first week and second week of training.
  Self Rate of Perceived Exertion (RPE) will be assessed via OMNI RES Scale (0-10 values) during resistance training (after every circuit) and 15-20 minutes after finishing each session.
Perception of Effort during Endurance Training. | Differences between first week and second week of training
  Borg Scale (6-20) will be used to collect the perception of effort during endurance training (every 5 minutes) and 15-20 minutes after each session.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Puente, Principal Investigator — University of Greenwich
Locations (1):
- University of Greenwich, Avery Hill Campus, Sparrows Farm. Avery Hill, London., United Kingdom, SE9 2BT, London, Avery Hill, London., United Kingdom

IPD SHARING:
Plan to Share IPD: No